CLINICAL TRIAL: NCT00100984
Title: A 48 Week Study Comparing Treatment With Saquinavir + Lopinavir/Ritonavir in Combination With Enfuvirtide HAART Versus Saquinavir + Lopinavir/Ritonavir + Other Nucleoside Combinations to See the Efficacy of These Treatments in Patients Infected With HIV-1
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: ML18021
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2005-12

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

INTERVENTIONS:
Drug: FUZEON [enfuvirtide]

SUMMARY:
The main objective of this study is to compare the safety and efficacy of an enfuvirtide containing regimen to a nucleoside combination regimen. Resistance information will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* CD4 cell count greater than 50 cells/mm^3
* HIV-1 RNA viral load greater than or equal to 5000 copies/mL
* Patients must be HIV treatment experienced
* Patients diagnosed with HIV-1 infection

Exclusion Criteria:

* Female patients must not be able to have children or must be under effective contraceptives
* Female patients who are pregnant
* Have taken enfuvirtide and/or T-1249 before
* Have serious kidney problems
* Alcohol and/or drug abuse
* Have had an organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-07-21 (Actual); Primary Completion 2005-07-16 (Actual); Study Completion 2005-07-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Hobson City, Alabama
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Atlanta, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Jackson, Mississippi
  - St Louis, Missouri
  - Newark, New Jersey
  - New York, New York
  - Huntersville, North Carolina
  - Dallas, Texas
  - Houston, Texas